CLINICAL TRIAL: NCT02163798
Title: Evaluation of Energy Expenditure and Cardiovascular Health Effects From Tai Chi and Walking Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Stanley Sai-Chuen Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHSRF 02030511
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Physical Activity
Keywords: Tai Chi; Walking; Physical activity; Randomized controlled trial; Chinese population; Exercise; Body composition; Cardiovascular risk factor; Energy expenditure; Fitness; SF-12
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tai Chi Group (Experimental): Participants in this group received a 12-week instructor-led Tai Chi training program.
  Interventions: Behavioral: 12-week instructor-led Tai Chi training program
- Walking Group (Experimental): Participants in this group received a 12-week instructor-led brisk walking training program.
  Interventions: Behavioral: 12-week instructor-led brisk walking training program
- Control Group (No Intervention): Participants in the control group did not receive intervention during the 12 weeks, and were told that they would be provided two sessions of free health and fitness evaluation with an interval of three months (12 weeks).

INTERVENTIONS:
Behavioral: 12-week instructor-led Tai Chi training program — A 12-week (45 min per day, 5 days per week) instructor-led Tai Chi training program was conducted in the Tai Chi group. Of the 5 days of exercise, 3 days were led by qualified instructors, and 2 other days for self-practice. Each session consisted of a 10-min standard warm-up, 30-min of Tai Chi exercise, and 5-min cool down stretching. The modified 32 Yang-style Tai Chi Chuan was used, because it could be learned within a relatively short time, and has been widely promoted in HK community. An exercise log was used to record the actual implementation of the training (instructor-led & self-practice).
  Arms: Tai Chi Group
Behavioral: 12-week instructor-led brisk walking training program — A 12-week (45 min per day, 5 days per week) instructor-led brisk walking training program was conducted in the walking group. Of the 5 days of exercise, 3 days were led by qualified instructors, and 2 other days for self-practice. Each session consisted of a 10-min standard warm-up, 30-min of walking exercise, and 5-min cool down stretching. An exercise log was used to record the actual implementation of the training (instructor-led & self-practice).
  Arms: Walking Group

SUMMARY:
Cardiovascular diseases (CVD) accounted for major mortality and morbidity rates in Hong Kong (HK) other than cancer. Increasing energy expenditure through regular exercise participation has been found to lower the risk of CVD such as hyperlipidemia and obesity. Healthcare professionals often prescribe lifestyle exercises for disease prevention, rehabilitation, and health maintenance purposes. Previous study revealed that Tai Chi and walking were widely practice by HK citizens. However, limited studies are found to compare the health benefits between Tai Chi and walking. Do Tai Chi and walking have equally effective in raising metabolic rate and reducing CVD risks? The difference in energy cost between a single bout of Tai Chi and walking has not been documented. Limited studies report the effects of Tai Chi in lowering the CVD risk. Since walking and Tai Chi are being heavily promoted in HK in recent years, there is an urgent need to document the evidence of these two common forms of exercise in terms of reducing CVD risks. Therefore, the purpose of the present study was to investigate the energy costs as well as CV health benefits, in terms of aerobic fitness, body composition, blood pressure, and blood lipid profiles, from the walking and Tai Chi exercise in a sample of HK Chinese adults, and to compare the effects between these two exercises. The investigators hypothesized that Tai Chi and walking had similar effects on improving energy cost and reducing CVD risks.

DETAILED DESCRIPTION:
An influential medical report released in 1996 confirmed that daily accumulation of 30 minutes of moderate physical activity would significantly lower the risks of many chronic diseases (Physical Activity and Health: A Report of the Surgeon General. Atlanta, GA: U.S. 1996). The report also recommended walking as one of the best forms of exercise that suitable for both healthy and patient population in all ages. To meet the daily 30 minutes exercise guidelines, a popular health promotion campaign -- 10,000 steps of walking per day, has been widely implemented in western countries, and has been recently promoted by the Health Info-World of HK Hospital Authority. Some studies demonstrated various health benefits from regular walking. The most recent study by Murphy et al. (Med Sci Sports Exerc. 2002) provided an excellent example that, in a 6-week walking program (5 days per week), one single bout of continuous 30 minutes of walking per day yielded similar health benefits as three 10-minute walks per day. The exercise intensity for both walking exercises was 70-80% of maximal heart rate, and resulted in significant increase in HDL-cholesterol, and decreases in triglycerides and total cholesterol. Both walking exercises improved body composition significantly. Moreover, tension/anxiety were also decreases significantly. Similar health benefits were also noted by several other studies (Moreau KL, et al. Med Sci Sports Exerc 2001. Wullink M et al. Med Sci Sports Exerc 2001. O'Hara RB et al. ACSM's Health Fitness J 2000). In these studies, the walking intervention periods varied from 6 weeks to 24 weeks, and daily walking times varied from 20 minutes to 50 minutes. Exercise intensities varied from 50% to 70% of VO2max. However, the energy cost of a typical walking bout of HK adults is not clear. Since body composition of HK Chinese is different from those reported for westerners, it is reasonably believe that the energy expenditure of walking for HK Chinese is different from those found in the literature. The CVD benefits result from walking have not been reported for the Chinese population. These outcome measures derived from walking and Tai Chi have not been compared.

Tai Chi is an ancient form of Chinese fitness exercise. A number of studies have investigated the positive health improvement effects from Tai Chi for patients (Channer KS et al. Postgrad Med J 1996. Fontana JA et al. Nurs Clin North Am 2000. Lan C et al. Med Sci Sports Exerc 1999), as well as for healthy individuals (Lan C et al. Med Sci Sports Exerc 1998. Zhuo D et al. Can J Appl sport Sci 1984). These health benefits include an improvement of aerobic fitness (Lai JS et al. J Am Geriatr Soc 1995. Hong YL et al. Br J Sport Med 2000) and energy metabolism (Zhuo D et al. Can J Appl sport Sci 1984. Schneider D et al. Int J Sport Med 1991), muscular strength and balance (Hong YL et al. Br J Sport Med 2000. Chan WW et al. Phys Occup Ther Geriatr 2000. Schaller KJ et al. J Gerontol Nurs 1996), as well as mental control (Jin P. J Psycho-som Res 1992. Fasko Jr D et al. Clin Kinesiol 2001). Compared to walking, it is intuitively perceived that Tai Chi is characterized by lower exercise intensity and metabolic cost. But surprisingly, Lan et al. reported that the exercise intensity of a typical session of Tai Chi (24 minutes Yang style) exceeded 70% of maximal heart rate (Lan C et al. Arch Phys Med Rehabil 1996). However, the energy cost of this single bout of Tai Chi has not been investigated. Tai Chi and walking seem to provide similar benefits but has not been compared simultaneously except in one study. Jin reported that heart rate, blood pressure, and urinary catecholamine changes for Tai Chi were similar to walking at a speed of 6 km/h (Jin P. J Psycho-som Res 1992). However, the energy cost and CVD risk measures were not investigated in this study. Although both walking and Tai Chi are believe to have positive health benefits, the extents to which these exercises contribute to raising the energy metabolism as well as CV health improvement have not been documented. Which form of exercise would elicit higher energy demand and produce greater CV health effects? Currently no scientific data available to report such results for HK Chinese. Results from this study will be valuable for practitioners to provide quantifiable prescriptions for obese individuals for weight control, as well as for those who need to improve CV health.

AIMS

Increasing energy expenditure has been considered a crucial role for reducing obesity. Raising the level of energy expenditure has also been found to produce improvement in cardio-respiratory fitness and lowering CVD risks. However, the energy cost from Tai Chi and walking have not been fully studied and their training effects on CVD risks have not been compared. The purpose of the present study was to examine the level of energy expenditure of Tai Chi and walking, and to compare the training effects from Tai Chi and walking in terms of lowering CVD risks. Specific aims of the project were as follows:

1. To evaluate the changes of energy expenditure, aerobic fitness, body composition, SF-12, blood serum lipid profiles (total, LDL, and HDL-cholesterols), fasting blood glucose, dietary habits and physical fitness after the 12 weeks of Tai Chi and walking training, respectively.
2. to compare the effects of Tai Chi and walking exercises on improving energy expenditure, aerobic fitness, body composition, SF-12, blood serum lipid profiles (total, LDL, and HDL-cholesterols), fasting blood glucose, dietary habits and physical fitness after the 12 weeks of Tai Chi and walking training.
3. compare the energy metabolism during these two exercises at similar practice intensity (approximately at 50-70% of age-predicted maximal heart rate, and 30 minutes of exercise bout).

ELIGIBILITY:
Inclusion Criteria:

* residents of large housing estates in the Shatin district
* physical inactivity
* no exercise habits

Exclusion Criteria:

* cardiovascular diseases
* pulmonary diseases
* neurological disorder
* musculoskeletal disorder

Ages: 36 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Changes of aerobic fitness after intervention | Measures were done at two time points: baseline and 3 months
  The aerobic fitness, in terms of maximal oxygen intake (VO2max in ml/min/kg), was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention VO2max minus the post-intervention VO2max was the "Changes of aerobic fitness after intervention"
Changes of resting VO2 (ml/min/kg) after intervention | Measures were done at two time points: baseline and 3 months
  Resting VO2 (ml/min/kg) was an indicator of resting energy expenditure (REE) in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention REE-VO2 minus the post-intervention REE-VO2 was the "Changes of resting VO2 after intervention"
Changes of body mass index (BMI) after intervention | Measures were done at two time points: baseline and 3 months
  BMI was an indicator of body composition in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention BMI minus the post-intervention BMI was the "Changes of BMI after intervention"
Changes of waist circumference (WC) after intervention | Measures were done at two time points: baseline and 3 months
  WC was an indicator of body composition in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention WC minus the post-intervention WC was the "Changes of WC after intervention"

SECONDARY OUTCOMES:
Changes of resting heart rate (HR in beats/min) after intervention | Measures were done at two time points: baseline and 3 months
  Resting heart rate (HR in beats/min) was an indicator of resting energy expenditure (REE) in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention REE-HR minus the post-intervention REE-HR was the "Changes of resting HR after intervention"
Changes of resting kilocalorie expenditure (KCal in KCal/min) after intervention | Measures were done at two time points: baseline and 3 months
  Resting KCal (KCal/min) was an indicator of resting energy expenditure (REE) in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention REE-KCal minus the post-intervention REE-KCal was the "Changes of resting Kilocalorie expenditure after intervention"
Changes of hip circumference (HC) after intervention | Measures were done at two time points: baseline and 3 months
  HC was an indicator of body composition in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention HC minus the post-intervention HC was the "Changes of HC after intervention"
Changes of waist hip ratio (WHR) after intervention | Measures were done at two time points: baseline and 3 months
  WHR was an indicator of body composition in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The pre-intervention WHR minus the post-intervention WHR was the "Changes of WHR after intervention"
Changes of body fat percentage after intervention | Measures were done at two time points: baseline and 3 months
  Body fat percentage was an indicator of body composition in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention body fat percentage minus the pre-intervention body fat percentage was the "Changes of body fat percentage after intervention"
Changes of skinfold thickness after intervention | Measures were done at two time points: baseline and 3 months
  Skinfold thickness was an indicator of body composition in our study. The sum of skinfold thickness was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention body fat percentage minus the pre-intervention body fat percentage was the "Changes of skinfold thickness after intervention"
Changes of SF-12 score after intervention | Measures were done at two time points: baseline and 3 months
  SF-12 score was an indicator of self-perceived health in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention SF-12 score minus the pre-intervention SF-12 score was the "Changes of SF-12 score after intervention"
Changes of blood pressure (BP) after intervention | Measures were done at two time points: baseline and 3 months
  Blood pressure was an indicator of cardiovascular health in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention BP minus the pre-intervention BP was the "Changes of BP after intervention"
Changes of fasting blood glucose (mmol/L) after intervention | Measures were done at two time points: baseline and 3 months
  Fasting blood glucose (mmol/L) was an indicator of cardiovascular health in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention fasting blood glucose minus the pre-intervention fasting blood glucose was the "Changes of fasting blood glucose after intervention"
Changes of total cholesterol (mmol/L) after intervention | Measures were done at two time points: baseline and 3 months
  Total cholesterol (mmol/L) was an indicator of cardiovascular health in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention total cholesterol minus the pre-intervention total cholesterol was the "Changes of total cholesterol after intervention"
Changes of high-density lipoprotein (HDL in mmol/L) after intervention | Measures were done at two time points: baseline and 3 months
  High-density lipoprotein (HDL in mmol/L) was an indicator of cardiovascular health in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention HDL minus the pre-intervention HDL was the "Changes of HDL after intervention"
Changes of Low-density lipoprotein (LDL in mmol/L) after intervention | Measures were done at two time points: baseline and 3 months
  Low-density lipoprotein (LDL in mmol/L) was an indicator of cardiovascular health in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention LDL minus the pre-intervention LDL was the "Changes of LDL after intervention"
Changes of triglycerides (mmol/L) after intervention | Measures were done at two time points: baseline and 3 months
  Triglycerides (mmol/L) was an indicator of cardiovascular health in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention triglycerides minus the pre-intervention triglycerides was the "Changes of triglycerides after intervention"
Changes of dietary habits after intervention | Measures were done at two time points: baseline and 3 months
  Dietary habits was measured by food frequency questionnaire (FFQ). It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The differences of two measurements were analyzed.
Changes of handgrip (kg) after intervention | Measures were done at two time points: baseline and 3 months
  Handgrip (kg) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention handgrip minus the pre-intervention handgrip was the "Changes of handgrip after intervention"
Changes of arm lift (kg) after intervention | Measures were done at two time points: baseline and 3 months
  Arm lift (kg) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention arm lift minus the pre-intervention arm lift was the "Changes of arm lift after intervention"
Changes of shoulder lift (kg) after intervention | Measures were done at two time points: baseline and 3 months
  Shoulder lift (kg) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention shoulder lift minus the pre-intervention shoulder lift was the "Changes of shoulder lift after intervention"
Changes of leg lift (kg) after intervention | Measures were done at two time points: baseline and 3 months
  Leg lift (kg) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention leg lift minus the pre-intervention leg lift was the "Changes of leg lift after intervention"
Changes of back lift (kg) after intervention | Measures were done at two time points: baseline and 3 months
  Back lift (kg) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention back lift minus the pre-intervention back lift was the "Changes of back lift after intervention"
Changes of balance test (sec) after intervention | Measures were done at two time points: baseline and 3 months
  Balance test (sec) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention balance test minus the pre-intervention balance test was the "Changes of balance test (sec) after intervention"
Changes of curl-up test (reps) after intervention | Measures were done at two time points: baseline and 3 months
  Curl-up test (reps) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention curl-up test (reps) minus the pre-intervention curl-up test (reps) was the "Changes of curl-up test (reps) after intervention"
Changes of sit-and-reach (leg, cm) after intervention | Measures were done at two time points: baseline and 3 months
  Sit-and-reach (leg, cm) was an indicator of physical fitness in our study. It was measured at baseline (pre-intervention) and 3 months (post-intervention), respectively. The post-intervention sit-and-reach (leg, cm) minus the pre-intervention sit-and-reach (leg, cm) was the "Changes of sit-and-reach (leg, cm) after intervention"
Six-month maintenance | 6-month after the completion of the training sessions
  To evaluate the adherence of the Tai Chi and walking exercise training, a questionnaire was administered at 6-month upon the completion of the training sessions to evaluate the maintenance situation of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Sai-Chuen Hui, EdD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong